CLINICAL TRIAL: NCT06113068
Title: Radiofrequency Using the Fistura® Procedure for the Treatment of Complex Anal Fistulas: Assessing Healing Rate and Anal Incontinence Up to 1 Year Follow-up
Brief Title: Fistura® Procedure for the Treatment of Complex Anal Fistulas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: F Care Systems NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fistura; NCT05899569 (obsolete NCT alias)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Complex Anal Fistulas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fistura procedure (Experimental)
  Interventions: Device: Fistura® procedure

INTERVENTIONS:
Device: Fistura® procedure — The Fistura® procedure is performed using a sterile Fistura® catheter (F Care Systems), intended to be connected to an F Care Systems radiofrequency generator (MedRF4000®). The flexible Fistura® catheters used during the procedure allow it to follow the path of the anal fistula, facilitating the closure of the fistula along its entire length. As the catheter can treat fistulas involving the sphincter complex, but without cutting or damaging it, it is expected to be effective in term of continence maintenance.

SUMMARY:
This study aims to evaluate the healing rate of complex fistulas using radiofrequency (Fistura® procedure), in a prospective, interventional, monocenter, single-arm design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with complex fistulas

   Complex fistulas include trans-sphincteric fistulas involving more than 30% of the external sphincter, supra-sphincteric fistulas, extra-sphincteric fistulas, horseshoe fistulas, fistulas involving multiple tracts (according to the ASCRS) and fistulas with a curved tract or a tract presenting diverticula, for which:

   Suppuration is described by the patient and/or visible by an opening in the anal margin or by anoscopy Clinical symptoms led to an MRI demonstrating the path Fistula path demonstrated in the acute phase during drainage of an abscess
2. Patient ≥ 18 years at study entry
3. Patients with a previously drained fistula, without diverticula > 10 mm, without T2 hyperintensity (assessed by MRI). Drainage is achieved by placing a seton, usually from 10 weeks to 12 months prior to the procedure
4. Patient and investigator signed and dated the informed consent form prior to the procedure

Exclusion Criteria:

1. Patient < 18 years at study entry
2. Patient has a known contraindication to treatment using radiofrequency (infectious anal pathologies, anal fissures, residual Longo anterior treatment staples)
3. Patient has a known contraindication to MRI
4. Simple fistulas defined as inter-sphincteric or trans-sphincteric, involving less than 30% of the total height of the sphincter apparatus (attested by MRI, ASCRS classification)
5. Patient has a fistula associated with radiation and inflammatory bowel disease
6. Patient is unable/unwilling to provide informed consent
7. Patient is unable to comply with the protocol or proposed follow-up visits and questionnaires
8. Patient is currently participating in another clinical study
9. Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Healing rate, clinically and MRI-assessed, at 12 months during an in-hospital visit | 12 months
  MRI-assessed healing (deep healing) is defined as a fibrous tract, a scarred tract, or a tract that is not visible on MRI. If the tract is shown to be inflammatory, liquid, or showing presence of diverticula, healing is considered to be not achieved.
  Clinical healing is defined as closure of the internal and external openings without inflammation or discharge or symptoms. Internal opening closure is confirmed by the absence of discharge and external opening closure is confirmed by visual and digital examination.

SECONDARY OUTCOMES:
Healing rate per type of fistulas treated | 12 months
  Include trans-sphincteric fistulas involving more than 30% of the external sphincter, supra-sphincteric fistulas, extra-sphincteric fistulas, horseshoe fistulas or fistulas involving multiple tracts
Anal incontinence at 2 weeks, and 2, 6 and 12 months | 2 weeks, 2 months, 6 months, 12 months
  Measured by the standard index of Jorge and Wexner
Healing rate without anal incontinence at 12 months | 12 months
Mean amount of energy used per treatment | At procedure
Duration of the procedure | At procedure
Return to daily activities at 2 weeks | 2 weeks
Return to work at 2 weeks | 2 weeks
Quality of life at 2 weeks, and 2, 6 and 12 months | 2 weeks, 2 months, 6 months, 12 months
  Measured by Quality of Life Anal Fistula Questionnaire (QoLAF-Q)
Rate and nature of late and immediate postoperative complications | At procedure, 2 weeks, 2 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHIREC site Braine l'Alleud-Waterloo, Braine-l'Alleud, Belgium

IPD SHARING:
Plan to Share IPD: No